CLINICAL TRIAL: NCT03102437
Title: FIX-HF-5CA: Continued Access Protocol for the Evaluation of the OPTIMIZER Smart System in Subjects With Moderate-to-Severe Heart Failure With Ejection Fraction Between 25% and 45%
Brief Title: Continued Access Protocol for the Evaluation of the OPTIMIZER Smart System
Acronym: FIX-HF-5CA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary objective of the protocol was to allow ongoing access to treatment of patients suffering from moderate to severe heart failure at selected investigational sites until the PMA was approved by the FDA for the OPTIMIZER System.
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP OPT2017-004
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure; Congestive Heart Failure; Chronic Heart Disease; CHF
Keywords: Cardiac Contractility Modulation; CCM; FIX-HF-5CA; Continued Access
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Continued Access
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Optimizer Smart System (Experimental): All eligible subjects will have the Optimizer Smart System implanted and receive cardiac contractility modulation therapy (CCM).
  Interventions: Device: Optimizer Smart System

INTERVENTIONS:
Device: Optimizer Smart System — The Optimizer Smart System delivers non-excitatory cardiac contractility modulating (CCM) electrical signals to the heart muscle. Treatment group subjects receive five non-contiguous one-hour periods of CCM signals per day.

SUMMARY:
This is a multicenter, prospective, single-arm Continued Access study of the Optimizer Smart System with CCM therapy.

DETAILED DESCRIPTION:
The Continued Access study is a prospective, non-randomized, multi-center study designed to allow controlled access to the Optimizer Smart System until the PMA order has been issued by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are 18 years of age or older
2. Subjects who have a baseline ejection fraction greater than or equal to 25% and less than or equal to 45% by echocardiography.
3. Subjects who, in the opinion of the Investigator (based on the current guidelines for clinical practice), have been treated for heart failure for at least 90 days and are currently receiving appropriate, stable medical therapy during the 30 days prior to enrollment for treatment of heart failure.
4. Subjects who are in New York Heart Association functional Class III and IV at the time of enrollment.
5. Subjects who are willing and able to return for all follow-up visits.

Exclusion Criteria:

1. Subjects who have a potentially correctible cause of heart failure, such as valvular heart disease or congenital heart disease.
2. Subjects receiving any form of inotropic support within 30 days before enrollment, including subjects on continuous IV inotrope therapy.
3. Subjects hospitalized for decompensated heart failure requiring acute treatment with intravenous loop diuretics, IV inotropes or hemofiltration within 30 days before enrollment and baseline testing.
4. Subjects who have a clinically significant amount of ambient ectopy, defined as more than 8,900 PVCs per 24 hours on baseline Holter monitoring.
5. Subjects having a PR interval greater than 375ms.
6. Subjects who are scheduled for a CABG or a PTCA procedure, or who have undergone a CABG procedure within 90 days or a PTCA procedure within 30 days of enrollment.
7. Subjects who have a biventricular pacing system, an accepted indication for such a device, or a QRS width of 130ms or greater.
8. Subjects who have had a myocardial infarction within 90 days of enrollment.
9. Subjects who have mechanical tricuspid valve.
10. Subjects who have a Left Ventricular Assist Device or prior heart transplant.
11. Subjects on dialysis.
12. Subjects who are participating in another experimental protocol.
13. Subjects who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Burkhoff, MD, PhD, Study Director — Impulse Dynamics
Locations (17):
- United States (17):
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - Southwest Cardiology Associates, Mesa, Arizona
  - Cardiovascular Consultants, Phoenix, Arizona
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Pima Heart, Tucson, Arizona
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Cooper University Hospital, Camden, New Jersey
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - St. Mary Research Institute, Langhorne, Pennsylvania
  - Jefferson Heart Institute, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Guthrie Medical Group at Robert Packer Hospital, Sayre, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - CHRISTUS Trinity Mother Frances Health System, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Optimizer Smart System (3-Lead): All eligible subjects will have the Optimizer Smart System 3-Lead implanted and receive cardiac contractility modulation therapy (CCM).
  Optimizer Smart System: The Optimizer Smart System delivers non-excitatory cardiac contractility modulating (CCM) electrical signals to the heart muscle. Treatment group subjects receive five non-contiguous one-hour periods of CCM signals per day.
- Optimizer Smart System (2-Lead): All eligible subjects will have the Optimizer Smart System 2-Lead implanted and receive cardiac contractility modulation therapy (CCM).
  Optimizer Smart System: The Optimizer Smart System delivers non-excitatory cardiac contractility modulating (CCM) electrical signals to the heart muscle. Treatment group subjects receive five non-contiguous one-hour periods of CCM signals per day.
Period: Overall Study
Arm/Group | Optimizer Smart System (3-Lead) | Optimizer Smart System (2-Lead)
Started | 70 | 36
Completed | 65 | 36
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimizer Smart System (3-Lead) | Optimizer Smart System (2-Lead) | Total
Number analyzed (Participants) | 70 | 36 | 106
Age, Continuous [Mean (Full Range); unit: years] | 65 [31 to 91] | 66 [33 to 84] | 66 [31 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 36
  Male | 44 | 26 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 59 | 30 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 36 | 106

OUTCOME MEASURES:

1. Primary Outcome: Observed Mortality Comparison to the Predicted Probability of Mortality
Description: The FIX-HF-5CA Study was unofficially intended to serve as the Post-Approval Study (PAS) with the intention of collecting 3 year observed mortality data and comparing that to the predicted probability of mortality derived from two validated heart failure models [MAGGIC (Meta-Analysis Global Group in Chronic Heart Failure) and SHFM (Seattle Heart Failure Model)]. The objective was to show that the observed prevalence of mortality was not worse than the derived predicted probability of mortality. Upon PMA and PMA Supplement approval of the device, however, FDA and the Sponsor stopped this 5CA study and a new PAS was initiated (NCT03970343). No long-term mortality data or final analysis was collected for this study.
Time Frame: 2 years 6 months
Population: All subjects implanted with the Optimizer System.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimizer Smart System (3-Lead) | Optimizer Smart System (2-Lead)
Number analyzed (Participants) | 70 | 36
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | Optimizer Smart System (3-Lead) | Optimizer Smart System (2-Lead)
All-Cause Mortality (participants affected / at risk) | 5/70 | 0/36
Serious Adverse Events (participants affected / at risk) | 13/70 | 4/36
Other Adverse Events (participants affected / at risk) | 12/70 | 3/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimizer Smart System (3-Lead) (N=70) | Optimizer Smart System (2-Lead) (N=36)
Optimizer Lead dislodgement (Surgical and medical procedures) | 2 (3) | 2 (2)
Optimizer Pocket infection (Infections and infestations) | 1 (1) | 0 (0)
Localized Infection (Infections and infestations) | 1 (1) | 0 (0)
ICD or pacemaker System AE (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmias (Cardiac disorders) | 2 (2) | 0 (0)
General Medical (General disorders) | 2 (2) | 0 (0)
General Cardiopulmonary event (Cardiac disorders) | 2 (2) | 1 (1)
Neurologic Dysfunction - TIA (Nervous system disorders) | 1 (1) | 1 (1)
Worsening Heart Failure (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimizer Smart System (3-Lead) (N=70) | Optimizer Smart System (2-Lead) (N=36)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
General Cardiopulmonary Event (Cardiac disorders) | 1 (1) | 1 (1)
Thromboembolism (non-Neurologic) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OPTIMIZER pocket stimulation (Surgical and medical procedures) | 1 (1) | 0 (0)
ICD inappropriate therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
General Medical (General disorders) | 8 (9) | 1 (1)

LIMITATIONS AND CAVEATS:
The FIX-HF-5CA Study was unofficially intended to serve as the Post-Approval Study (PAS) with the intention of collecting 3 year data. Upon PMA (3-lead) and PMA Supplement approval (2-lead) of the device, however, FDA and the Sponsor terminated this continued access study and a new PAS was initiated (NCT03970343). No long-term or final analysis was collected for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Publication Committee shall consist of the National PIs and Impulse Dynamics representatives. All abstracts and papers of the multi-center publications will be reviewed by members of the publication committee and all authors. When appropriate, the publication committee will collect comments and resolve final draft issues. If a paper is rejected, the publication committee and its authors will decide the next course of action.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT03102437/Prot_ICF_001.pdf